CLINICAL TRIAL: NCT06168435
Title: e-IMPAQc Implementation and Evaluation of a Mobile Application for the Systematic Assessment of Patient and Caregiver Reported Outcomes in Quebec Across the Cancer Continuum (eIMPAQc)
Brief Title: e-IMPAQc Systematic Assessment of Patient Reported Outcomes in Cancer Care
Acronym: eIMPAQc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: St. Mary's Research Center, Canada (Other)
Responsible Party: Principal Investigator, Sylvie Lambert, Principal Scientist, St. Mary's Research Center, Canada
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: SMHC 18-24
Record Dates: First submitted 2023-08-14; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: ePRO
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation (No Intervention): Outcomes collected in patient populations prior to roll-out of the eIMPAQc
- Post-implementation (Experimental): Outcomes collected in patient populations after roll-out of eIMPAQc
  Interventions: Other: eIMPAQc

INTERVENTIONS:
Other: eIMPAQc — e-IMPAQc has five main components: 1) primary and secondary standardized e-PRO questionnaires and algorithm; 2) summary report for clinicians with alert system; 3) summary report for patients, with tailored notifications regarding symptom severity; 4) self-management fact sheets library; and 5) clinical dashboard.
  Arms: Post-implementation

SUMMARY:
Purpose: The Electronic Implementation of Patient and Caregiver Reported Outcomes across cancer centres in Quebec project, or e-IMPAQc, was launched in 2017. e-IMPAQc's goal is to actively engage patients, their caregivers, healthcare professionals (HCPs), managers, policy makers, researchers and IT personnel to co-develop, implement, and evaluate an evidence-informed electronic patient-reported outcomes (e-PRO) screening and management program across Quebec.

Methods: e-IMPAQc built on the Improving Patient Experience and Health Outcomes Collaborative (iPEHOC) project, the first initiative in the province to implement e-PRO screening and was rolled out in three phases. e-IMPAQc has five main components: 1) primary and secondary standardized e-PRO questionnaires and algorithm; 2) summary report for clinicians with alert system; 3) summary report for patients, with tailored notifications regarding symptom severity; 4) self-management fact sheets library; and 5) clinical dashboard. Phase 1 included initiating change management and the co-development of the e-PRO algorithm with patients, their caregivers, HCPs, managers, policy makers, researchers and IT personnel (herein collectively referred as stakeholders) across seven cancer centres. The iPEHOC algorithm was used as a starting point given its successful implementation in one of the participating cancer centres for several years. Phase 1 also included feasibility work to establish a caregiver-reported outcomes (CROs) algorithm as well as the identification and configuration of appropriate electronic platforms on which to house e-IMPAQc. In Phase 2 the focus was on preparing for imminent implementation through workflow mapping and putting in place implementation support (e.g., site coordinators). A pilot of e-IMPAQc (excluding CROs) was also undertaken at one of the participating centres. In Phase 3, e-IMPAQc is being sequentially rolled out to as many cancer centres as possible and then evaluated. Qualitative and quantitative methods are used to document the process of implementation, patient and caregiver, and knowledge transfer (KT) outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Receiving cancer care at designated center

Exclusion Criteria:

* Unable to speak English or French
* Unable to use email and internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom severity | Baseline, 4 months
  Symptom severity as measured by the population-specific eIMPAQc symptom screening algorithm, including the Edmonton Symptom Assessment System Revised (ESAS-r) screening measures. Severity is measured on a scale of 0-10.
Patient perception of communication with health care team | Baseline, 4 months
  6 item Clinician-patient communication subscale of the Primary Care Assessment Survey (PCAS), provides an overall score
Patient activation | Baseline, 4 months
  13 items Patient Activation Measure provides an overall score
Quality of life | Bsaseline,4 months
  The EQ-5D-5L is used to measure health related, quality of life. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each level is rated on scale that describes the degree of problems in that area.
Emergency room visits | In the 18 months following consent
  Using hospital administrative data, we will report on the number of individual visits to the emergency room
Survival | In the 18 months following consent
  Incidence of mortality
Feasibility of using the eIMPAQc ePRO system in cancer care centres | Throughout the implementation period, over the course of each participants' 4-6 month follow-up period
  Feasibility of using the eIMPAQc symptom screening and management program will be measured using the following metrics:
  * Rates of consent to use eIMPAQc among eligible patients referred/invited to patriciate
  * Rates of administration and completion of the eIMPAQc ePRO screening processes
  * Number and timing of withdrawals
  * Number of eIMPAQc ePRO screenings that generate an alert and/or clinical action
  Metrics will be combined with qualitative data from semi-structured interviews with participants to provide an overall assessment of feasibility
Acceptability of using the eIMPAQc ePRO system in cancer care centres | Throughout the implementation period, over the course of each participants' 4-6 month follow-up period
  Acceptability of the components of the eIMPAQc program will be assessed through a 40 item eIMPAQc acceptability questionnaire
Satisfaction | 4 months
  Measured using the 8 item Client Satisfaction Questionnaire (CSQ-8)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mary's Research Centre, Montreal, Quebec, Canada